CLINICAL TRIAL: NCT06704503
Title: To Study the Changes Under Different Accommodation of Anterior Eye in People of Different Ages and 3D Crystal Reconstruction.
Brief Title: The Changes Under Different Accommodation of Anterior Eye and 3D Crystal Reconstruction.
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0939
Record Dates: First submitted 2024-11-17; First posted 2024-11-26 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Accommodation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Age 20-80 years old; Astigmatism ≤-1.50D; Best corrected visual acuity ≥4.9. Excluding people with other systemic underlying diseases; Have a history of eye surgery; Patients with intraocular lens or aphakia; Patients with strabismus and amblyopia; Pregnant or lactating women; People with mental disorders or neurological diseases who cannot cooperate with the examination;
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A was 20-40 years old: They were divided into three groups according to age: A, B, and C.Group A was 20-40 years old.
- Group B was 40-60 years old: They were divided into three groups according to age: A, B, and C. Group B was 40-60 years old.
- Group C was 60-80 years old: They were divided into three groups according to age: A, B, and C. Group C was 60-80 years old.

SUMMARY:
Accommodation is defined as a dynamic change in the overall refractive power of the eye during near fixation. Despite extensive investigations, the exact nature of human accommodation remains controversial. And recent alternative theories question the original concept of accommodation.Different experts have put forward different hypotheses. The age-related changes that underlie presbyopia are also not fully understood.Because of these unanswered questions, the topic of regulation and presbyopia remains a focus of research.

DETAILED DESCRIPTION:
Accommodation is the process by which the eye changes the shape and diopter of the lens to obtain a clear image of an object at different distances. Despite extensive research on regulation, the exact nature of human regulation remains controversial. Age-related changes in presbyopia are also not fully understood. Some studies have shown that a hardening of the lens and an increase in the thickness and diameter of the lens with age can lead to presbyopia. Others believe that the main cause is external lens factors, such as age-related changes in the Angle of lens suspension ligament attachment, reduced ciliary body movement, etc. Due to these unanswered questions, the topic of regulation and presbyopia remains the focus of research. In living humans, modulation studies utilize different imaging modes, and ultrasound biomicroscopy (UBM) and Optical Coherence Tomography(OCT) are particularly important in studying anterior segments and modulation. However, UBM is a contact inspection and requires highly skilled technicians. And UBM cannot image the entire anterior segment in a single capture. Anterior segment OCT (AS-OCT), on the other hand, is non-invasive and provides higher resolution imaging, allowing us to capture the morphology of the anterior segment structures in different populations and the changes of the anterior segment structures in response to regulatory stimuli. Studies have shown that with age, reduced anterior chamber depth, pupil contraction, increased lens thickness, increased lens arch height, and loss of posterior ciliary muscle contraction may be biomarkers of early presbyopia. In this study, anterior segment OCT was used to explore whether there were differences in the structural morphology of the anterior segment in people of different ages, and what changes occurred in the structure of the anterior segment after initiation of regulation.

ELIGIBILITY:
Inclusion Criteria:

· Patients with astigmatism ≤-1.50D and best corrected visual acuity ≥4.9

Exclusion Criteria:

* Patients with other systemic diseases
* Patients with a history of eye surgery
* Patients with intraocular lens or aphakia
* Patients with strabismus and amblyopia
* Pregnant or lactating women
* People with mental disorders or neurological diseases who cannot cooperate with the examination

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age 20-80 years old; Astigmatism ≤-1.50D; Best corrected visual acuity ≥4.9;Excluding other systemic underlying diseases; Have a history of eye surgery; Patients with intraocular lens or aphakia; Patients with strabismus and amblyopia; Pregnant or lactating women; People with mental disorders or neurological diseases who cannot cooperate with the examination;
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Central corneal thickness changes during accommodation | Baseline, after accommodation(30 minutes after using pilocarpine)
  Central corneal thickness CCT(μm)
peripheral corneal thickness changes during accommodation | Baseline, after accommodation(30 minutes after using pilocarpine)
  peripheral corneal thickness(μm)
anterior chamber depth changes during accommodation | Baseline, after accommodation(30 minutes after using pilocarpine)
  anterior chamber depth ACD(mm)
anterior chamber Angle Angle changes during accommodation | Baseline, after accommodation(30 minutes after using pilocarpine)
  anterior chamber Angle Angle ACA(°)
anterior opening distance changes during accommodation | Baseline, after accommodation(30 minutes after using pilocarpine)
  anterior opening distance AOD(mm)
pupil size changes during accommodation | Baseline, after accommodation(30 minutes after using pilocarpine)
  pupil size PD(mm)
lens thickness changes during accommodation | Baseline, after accommodation(30 minutes after using pilocarpine)
  lens thickness LT(mm)
anterior and posterior surface curvature radius changes during accommodation | Baseline, after accommodation(30 minutes after using pilocarpine)
  anterior and posterior surface curvature radius(mm)
lens arch height changes during accommodation | Baseline, after accommodation(30 minutes after using pilocarpine)
  lens arch height LV(mm)
lens sagittal height changes during accommodation | Baseline, after accommodation(30 minutes after using pilocarpine)
  lens sagittal height(mm)
anterior chamber volume changes during accommodation | Baseline, after accommodation(30 minutes after using pilocarpine)
  anterior chamber volume(mm³)
posterior chamber volume changes during accommodation | Baseline, after accommodation(30 minutes after using pilocarpine)
  posterior chamber volume(mm³)
crystal equatorial diameter changes during accommodation | Baseline, after accommodation(30 minutes after using pilocarpine)
  crystal equatorial diameter(mm)

CONTACTS AND LOCATIONS:
Overall Officials: Wen Xu, Phd, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided